CLINICAL TRIAL: NCT05506501
Title: Comparative Study Between Intentional Unilateral Epidural Block Versus Ultrasound Guided Combined Femoro-sciatic Nerves Block for Patients With Low Ejection Fraction Undergoing Insertion of Nail Tibia for Fixation of Fracture Shaft Tibia
Brief Title: Unilateral Epidural Block Versus Ultrasound Guided Combined Femoro-sciatic Nerves Block for Patients With Low Ejection Fraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OFT IRB00006379
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Low Ejection Fraction Patients; Fracture Tibia
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral epidural anesthesia group (Active Comparator): Forty patients with low ejection fraction (30-40%) will do elective insertion of nail tibia for fixation of fracture shaft tibia using unilateral epidural anesthesia.
  Interventions: Procedure: unilateral epidural anesthesia
- Ultrasound guided femoro/ sciatic nerve block group (Active Comparator): Forty patients with low ejection fraction (30-40%) will do elective insertion of nail tibia for fixation of fracture shaft tibia by femoral/sciatic nerve block using ultrasound guidance.
  Interventions: Procedure: Ultrasound guided femoro/ sciatic nerve block

INTERVENTIONS:
Procedure: unilateral epidural anesthesia — Forty patients with low ejection fraction (30-40%) will do elective insertion of nail tibia for fixation of fracture shaft tibia using unilateral epidural anesthesia.
  Other Names: Ultrasound guided femoro/ sciatic nerve block
  Arms: Unilateral epidural anesthesia group
Procedure: Ultrasound guided femoro/ sciatic nerve block — Forty patients with low ejection fraction (30-40%) will do elective insertion of nail tibia for fixation of fracture shaft tibia by femoral/sciatic nerve block using ultrasound guidance.
  Arms: Ultrasound guided femoro/ sciatic nerve block group

SUMMARY:
compare unilateral epidural anesthesia versus femoral/sciatic nerve block by ultrasound guided as anesthetic technique for cases with low ejection fraction undergoing insertion of nail tibia for fixation of fracture shaft tibia.

DETAILED DESCRIPTION:
Group A ;( Unilateral epidural anesthesia group) Forty patients with low ejection fraction (30-40%) will do elective insertion of nail tibia for fixation of fracture shaft tibia using unilateral epidural anesthesia.

Group B;;( Ultrasound guided femoro/ sciatic nerve block group) Forty patients with low ejection fraction (30-40%) will do elective insertion of nail tibia for fixation of fracture shaft tibia by femoral/sciatic nerve block using ultrasound guidance.

For each patient, onset of sensory and motor block, degree of motor block, sign of sensory block in the contralateral lower limb for the epidural group, success in providing adequate anesthesia, hemodynamic changes, time of first analgesic request will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years old.
* Patients scheduled for elective insertion of nail tibia for fixation of fracture shaft tibia.
* Patients with low ejection fraction (30-40%).

Exclusion Criteria:

* Patient refusal
* Uncooperative patient
* Unconscious patients
* Cases with head trauma
* History of relevant drug allergy to local anesthetics
* Local infection at the site of the block
* Patients with coagulopathies and impaired platelet functions
* Patients with hemodynamic instability
* Previous neurological deficit in lower limb and previous femoral artery grafts or injuries.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
mean blood pressure | 20 minutes after anesthesia

SECONDARY OUTCOMES:
adequate sensory block | 20 minutes after the block
adequate motor block | 15 minutes after the block
time of first analgesic request | within 24 hours after the block

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes